CLINICAL TRIAL: NCT01831180
Title: A Comparison of Scalp Blood Flow and Hair Shaft In Premenopausal Women Versus Postmenopausal Women: II-Scalp & Blood Flow 2012
Brief Title: A Comparison of Scalp Blood Flow and Hair Shaft In Premenopausal Women Versus Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00022675
Record Dates: First submitted 2013-04-02; First posted 2013-04-15 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: hair; scalp; blood flow; Caucasian; Histamine stimulation; Wake Forest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Premenopausal women 19-25 yrs
- Postmenopausal 60 yrs +

SUMMARY:
The purpose of this study is to compare the differences in various chemical and biologic parameters of scalp and and hair parameters between young and old Caucasian females. The hair state and scalp blood flow in younger and older age groups with typical hair care practices will be qualified by measuring various parameters of the hair shaft and scalp with correlation back to hair and scalp satisfaction as measured in the subject. This is a single center study with an anticipated 4 month enrollment period. The investigators will compare various scalp and hair parameters between young and old Caucasian females by obtaining the following biological and chemical/structural information. Hair growth rate, anagen to telogen ratio, hair density (determined via phototrichogram and digital imaging), Vascular blood flow (Laser Doppler Flowmetry), Histamine stimulation and Hair diameter (clipped hairs). In addition, a detailed questionnaire will be administered to each subject regarding satisfaction of the subject's hair state, including typical hair care regimens and symptoms in scalp and/or hair shafts. This information will be correlated to the biologic and chemical/structural information about hair and scalp health. Approximately 50 healthy, Caucasian female subjects will be enrolled in this study. Twenty five participants will be 19-25 years-old and 25 participants 60 years or older. There will be two visits, Baseline and approximately 48 hours after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to sign informed consent
* Female in age groups 19-25 years old and 60 years or older
* Must be of Caucasian descent, to avoid any ethnic differences in hair biology or pigment among different races
* Must be willing to have a thorough scalp and hair shaft examination
* Must be willing to discuss current and past hair care regimens
* Must have washed hair at least 48 hours, but not less than 12 hours prior to study visit
* Must be willing to not wash hair between Baseline and second visit.
* Pregnant and nursing females will not be allowed in the study; a baseline pregnancy test will be done to exclude pregnancy on females of childbearing potential
* Must be >6 months (26 weeks) postpartum
* Must have sufficient contrast between scalp skin color and hair color (Fitzpatrick skin type I-IV)
* Must have hair at least 2 inches long
* May have mild itching and mild scaling of the scalp, but not dandruff
* Must be willing to have hair clipped and shaved to 1 mm within an approximately 1cm2 test site
* Must be a non-smoker for the past 6 months
* Must be in good stable general health, with no current infections
* Must be able to return to the study site 48 hours after the Baseline visit for the second visit.

Exclusion Criteria:

* Must not have hypertension, diabetes, or any neurological disease since all these can affect scalp blood flow
* Must not take any antihistamines for two weeks prior to the baseline visit and throughout the study.
* Must not have any known allergy or past history of anaphylaxis to histamine
* May not have sewn-in or glued hair pieces or extensions at the time of the study
* Must not cut hair during the study
* Must not have hair loss beyond what is considered normal in the opinion of the Investigator at the time of the study
* Must not color hair or have other salon-type procedures (relaxer, permanent, highlighting, etc.) performed within 2 weeks of the initial visit
* Must not have any other underlying scalp disorder that could interfere with the test procedures or findings
* Must not have lost ≥10% of body weight within the past 12 months
* Must not have been on a weight reduction program overseen by a physician or nutritionist within the past 12 months
* Has used hair growth products e.g. minoxidil in the past 18 months
* Has undergone a hair transplant or scalp reduction surgery
* Has participated in a hair growth study within the past 15 months
* Is currently participating in another clinical study at this or any other facility
* Is taking, for a chronic condition, any prescription or over the counter medication(s) that in the opinion of the Investigator are likely to affect the hair properties (e.g. immunosuppressive agents, corticosteroids, or chronic use of anti-inflammatory medication)
* Application of any over-the-counter or prescription drug to the scalp on a routine basis within the past 3 months including but not limited to retinoids (e.g. retinal, tretinoin, retinylpalmitate, retinyl acetate, retinyl propionate), topical corticosteroids, benzyl peroxide, or any topical hormone therapy (e.g. Eterna 27)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Selected from the Wake Forest University Health Sciences Dermatology clinics and responders to Institutional Review Board (IRB) approved advertising
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Scalp/Hair Biological Structural | Baseline
  Two areas will be tested in total; one site on the scalp (parietal scalp: which is the area between top of the scalp and either ear) and one area on the forearm. Study staff will take a template and mark off the designated scalp area with a marker. This temporary ink mark will be used as a reference point. The hairs in the marked area (approximately the size of a nickel) will be cut and clipped to 1 millimeter in length for analysis. A digital photographic image of the scalp and hair shafts (phototrichogram) will be taken at the clipped hair site of the scalp. The temporary ink mark that was placed during hair cutting/clipping will be used as a reference point to position the image for capture and storage.
Scalp/Hair Biological Structural | 48 hours after baseline
  A site on the forearm will be marked as control on the second visit for laser blood flow measurements. Forearm and scalp blood flow will be assessed with Laser Doppler Imager (LDI) on the marked sites. Scalp reactive hyperemia (scalp blood flow) will be measured by injecting just under the skin a small amount of histamine (100 µg of histamine dihydrochloride in 1 ml normal saline) using small needle at both the chosen scalp and forearm sites. Then the blood flow measurement with the LDI will be repeated at the above mentioned sites 1 minute after histamine injection. The study staff will take another digital image (phototrichogram) of the clipped scalp area. The temporary ink mark placed during the baseline visit will serve as a reference point.

SECONDARY OUTCOMES:
Hair Chemical Structural information | Baseline
  Chemical/Structural information Hair diameter (clipped hairs: Hair fiber diameter will be measured on the recovered hair from the initial clipping site. The analysis will be completed at an external laboratory using the OFDA100 instrument.
  The OFDA100 method allows measurement of the hair diameter from all of the individual hairs in the sample - enabling analysis of the diversity of the population of hairs. This method enables looking at the overall diameter of the population in a single sample, comparing the number of modes, the proportion of each mode, and also the individual diameters and variability of each mode.
Hair Chemical Structure | 48 hours after baseline
  Chemical/Structural information Hair diameter (clipped hairs: Hair fiber diameter will be measured on the recovered hair from the initial clipping site. The analysis will be completed at an external laboratory using the OFDA100 instrument.
  The OFDA100 method allows measurement of the hair diameter from all of the individual hairs in the sample - enabling analysis of the diversity of the population of hairs. This method enables looking at the overall diameter of the population in a single sample, comparing the number of modes, the proportion of each mode, and also the individual diameters and variability of each mode.

OTHER OUTCOMES:
Scalp/Hair Care Practices | Baseline
  A self assessment questionnaire of hair type, care practices, attitudes, and beliefs.
Scalp/Hair Care Practices | 48 hours after baseline
  A follow-up self assessment questionnaire of hair type, care practices, attitudes, and beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine - Dermatology Clinic, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No